CLINICAL TRIAL: NCT02923154
Title: An Exploratory Study of MT-3995 in Patients With Non-Alcoholic Steatohepatitis(NASH) (Placebo-Controlled Double-Blind Study)
Brief Title: Efficacy and Safety of MT-3995 in Patients With Non-Alcoholic Steatohepatitis(NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-3995-J07
Record Dates: First submitted 2016-10-02; First posted 2016-10-04 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: NASH
Keywords: NASH
MeSH Terms: interventions — apararenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT-3995 (Experimental)
  Interventions: Drug: MT-3995
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-3995
  Arms: MT-3995
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, tolerability and pharmacokinetics of multiple oral administration of MT-3995 in patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with NASH before randomization
* Subjects who conducts diet or exercise therapy at the beginning of run in period.
* Subjects who has given full and adequate information of the protocol and with written informed consent

Exclusion Criteria:

* Subjects with hepatic failure or previously diagnosed with hepatic cirrhosis
* Subjects with alcohol dependence or previously diagnosed with alcohol dependence
* Subjects with other chronic liver disease (e.g., primary sclerosing cholangitis, alcoholic liver damage, hemochromatosis, Wilson's disease)
* Presence, history, or family history of long QT syndrome or Torsades de Pointes
* Subjects with heart failure (New York Heart Association Class III-IV)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in ALT | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in ALT | 24 weeks
Adverse events | From baseline to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (2):
- Japan (2):
  - Investigational site, Kanagawa
  - Investigational site, Osaka